CLINICAL TRIAL: NCT04558333
Title: CLAD: Finding Biomarkers to Predict Rejection and/ or Outcome After Lung Transplantation
Status: Terminated | Type: Observational
Why Stopped: lack of resources (personnel and budget)
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Therese Lapperre, Prof. Dr. Lapperre, University Hospital, Antwerp
Other Study IDs: CLAD
Record Dates: First submitted 2020-09-09; First posted 2020-09-22 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Lung Transplant Failure and Rejection; Primary Graft Dysfunction
MeSH Terms: conditions — Rejection, Psychology; Primary Graft Dysfunction | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the first 72 hours after transplantation cell free DNA will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LTx (lung transplant) patients: identification of possible biomarkers
  Interventions: Other: blood and exhaled breath specimens

INTERVENTIONS:
Other: blood and exhaled breath specimens — identification of possible biomarkers

SUMMARY:
Lung transplantation is the ultimate treatment for end stage lung diseases. Survival after lung transplantation is limited mainly due to the development of chronic allograft dysfunction (CLAD). Both acute cellular rejection and primary grade dysfunction (PGD) have been associated with the development of CLAD. In this study we will investigate multiple prognostic factors that influence long term survival after lung transplantation with a specific interest in PGD, acute rejection and the development of CLAD.

DETAILED DESCRIPTION:
At specific time points (according to protocol) exhaled breath, blood specimens, bronchoalveolar lavage and biopsies will be collected. These will be analyzed in an attempt to identify possible biomarkers that will predict the development of PGD and/or CLAD.

ELIGIBILITY:
Inclusion Criteria:

* all lung transplant recipients > 18 years signed ICF (informed consent form)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all lung transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
identify prognostic biomarkers in blood, bronchoalveolar lavage and exhaled breath that will determine long term survival after human lung transplantation. | up to 520 weeks
  death

SECONDARY OUTCOMES:
Secondary objectives are obtaining information on the development of (Primary graft development) PGD in relationship to respiratory viruses, genetic profile and exhaled breath in patients and (if possible donors) after human lung transplantation. | from transplantation till 72 hours after surgery
  PGD

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse Lapperre, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium